CLINICAL TRIAL: NCT03037671
Title: Evaluation of Malglycemia Via Continuous Glucose Monitoring in the Pediatric Hematopoietic Stem Cell Transplant Population
Brief Title: Evaluation of Malglycemia Via Continuous Glucose Monitoring in the Pediatric HSCT Population
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 16-2250.cc
Record Dates: First submitted 2017-01-25; First posted 2017-01-31 (Estimated); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Hematopoietic Stem Cell Transplantation
Keywords: Malglycemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CGM Monitored Cohort: The continuous glucose monitor (CGM) used during this study will be the Abbot Freestyle Libre Professional Continuous Glucose Monitoring System.
  Interventions: Device: Continuous Glucose Monitor (CGM)

INTERVENTIONS:
Device: Continuous Glucose Monitor (CGM) — Participants will wear the continuous glucose monitor (GCM) device during the peri-HSCT period for the duration of their initial hospital admission. No intervention based on results.
  Other Names: Abbot Freestyle Libre Pro

SUMMARY:
This study is designed to determine feasibility of using a continuous glucose monitor in pediatric, adolescent and young adult hematopoietic stem cell transplant (HSCT) recipients, and to identify the incidence and risk factors for malglycemia in primary admission for pediatric, adolescent and young adult HSCT patients as well as to characterize the relationship between outcomes and malglycemia in this population.

DETAILED DESCRIPTION:
This study is a prospective observational cohort analysis examining the rate of malglycemia in the pediatric HSCT population and the effect of malglycemia on important post-HSCT outcomes. In addition to usual care during the peri-HSCT period, participants in this trial will be asked to wear a continuous glucose monitor for the duration of their initial hospital admission. Participants will wear this monitor while admitted to the hospital for up to one week prior to transplant, and up to 60 days after transplant.

ELIGIBILITY:
Inclusion Criteria:

1. Patients age 2 to 30 years old at time of transplant.
2. Patients undergoing hematopoietic stem cell transplantation at CHCO.
3. Subject willing to wear a continuous glucose monitor for the duration of the study.
4. Subject willing to follow study protocols.

Exclusion Criteria:

1. Preexisting diagnosis of type 1 diabetes, type 2 diabetes, or an insulin requirement in the 2 weeks preceding transplant.
2. Preexisting condition requiring use of steroids (other than HSCT)
3. Severe psychiatric disease or developmental delays that might interfere with ability to provide informed consent.
4. Any other medical condition which in the opinion of the investigators impairs the person's ability to safely participate in the trial.
5. Subject has an active skin condition that would affect sensor placement.

Ages: 2 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This study will enroll 23-30 subjects undergoing hematopoietic stem cell transplant at Children's Hospital Colorado.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2017-02-09 (Actual); Primary Completion 2020-01-17 (Actual); Study Completion 2024-04-04 (Actual)

PRIMARY OUTCOMES:
The number of patients with Malgylcemia | 1 week prior to transplant through maximum 60 days post-transplant; inpatient only
  Hypoglycemia (BG < 70 mg/dL), hyperglycemia (BG ≥ 126 mg/dL), or glycemic variability (σ ≥ 29 mg/dL). Participants will wear a continous glucose monitor (CGM) to measure glycemia levels. This will service both as an exposure and and outcome.
The number patients that contract an infection | 0-100 days post-transplant
  Infection, defined by clinically significant positive microbiology or radiology result

SECONDARY OUTCOMES:
The length of hospital stays for all participants | Through study completion to 1 year of follow-up
  Days in the hospital post-transplant
The length of hospital stays in the ICU for all participants | Through study completion to 1 year of follow-up
  Number of days in the intensive care unit (ICU) during primary HSCT admission
The Graft-versus-host-disease (GVHD) status of all participants | Through study completion to 1 year of follow-up
  Graft-versus-host status and time to graft-versus-host will be analyzed

CONTACTS AND LOCATIONS:
Overall Officials: Jenna M Demedis, MD, Principal Investigator — Children's Hospital Colorado
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No